CLINICAL TRIAL: NCT00424697
Title: A Randomized, Placebo-controlled, Double-dummy, Four-way Crossover Design Study to Investigate the Changes of fMRI BOLD Activation Induced by Emotional Activation Paradigms Following Single Doses of GW876008 and Lorazepam (Comparator) in Healthy Subjects.
Brief Title: A Study to Investigate the Effects of GW876008 on Brain Activation During Emotional Processing in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CRH104150
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: Brain imaging,; fMRI,; stimulation,; pharmacodynamics,; tolerability,; healthy subjects
MeSH Terms: interventions — Lorazepam; GW 876008

INTERVENTIONS:
Drug: placebo
Drug: lorazepam
Drug: GW876008
  Other Names: placebo; lorazepam

SUMMARY:
Data suggests that imaging activity of the brain can measure the effects of anti-anxiety drugs. This study will investigate the effect of GW876008 on areas of the brain involved with thinking and emotion

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-50 years, inclusive.
* STAI-trait score = or > 40.
* STAI-state score <50th percentile of the normal population distribution.
* Female subjects of non-childbearing.
* Female subjects of childbearing potential must agree to use appropriate contraception.
* Healthy subjects, as determined by a responsible physician
* Body weight ≥ 50 kg (110 lbs), and BMI within the range 19-29.9 kg/m2 inclusive.
* Demonstrates no significant evidence of active disease, physical or mental impairment when assessed by qualified personnel
* Non-smoker (abstinence from smoking for at least 6 months before the start of the study).
* Normal electrocardiogram.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* Provide a signed and dated written informed consent prior to study participation

Exclusion Criteria:

* As a result of any of the medical interview, physical examination, evaluation of mental state and psychiatric history or screening investigations the physician responsible considers the subject unfit for the study.
* Any history of suicidal attempts or behaviour.
* Any history or current diagnosis of a psychiatric illness.
* Any history of an endocrine disorder including, but not limited to, diabetes or disorders of the hypothalamus, pituitary, adrenal, or thyroid glands, or gonadal disorder or dysfunction of the reproductive organs.
* Abnormal pepsinogen I level at screening.
* Liver Function Tests (LFTs) elevated above the reference range at pre-study screening that remain elevated with a repeat LFT
* Any other clinically significant laboratory abnormality.
* Positive faecal occult blood test.
* Positive pre-study urine drug/alcohol breath screen.
* Positive pre-study HIV 1/2, Hepatitis B surface antigen and positive Hepatitis C antibody result within 3 months of the start of the study.
* Pre-existing or current Helicobactor pylori infection.
* History of alcohol/drug abuse or dependence within 12 months of the study
* Consumption of grapefruit juice or grapefruit within 14 days prior to the first dose of study medication.
* History of peptic ulcer disease.
* Abnormal screening ECG
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* Systolic blood pressure < 90mmHg or >140mmHg; diastolic blood pressure < 60mmHg or > 90mmHg; pulse rate < 40bpm or > 90bpm.
* Participation in a clinical trial with a drug or new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History or current diagnosis of acute narrow angle glaucoma.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecystectomy) which would be expected to influence the absorption of drugs.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* Subjects who are left handed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Differences in brain activation elicited by Matching Emotional Face Expression paradigm following single oral doses of GW876008 and lorazepam on day 1, sessions 1-4

SECONDARY OUTCOMES:
GW876008 blood levels | pre-dose & post-dose, sessions 1-4
clinical rating scales change after dosing: questionnaires collected | pre-dose & up to 6-8 hours post-dose.
Safety: 12-lead ECG, vital signs, adverse events, clinical labs
fMRI BOLD neuroanatomical structure of the emotional brain neurocircuitry and connectivity
fMRI BOLD Signal characteristics and connectivity
fMRI BOLD Response in the emotional brain neurocircuitry and occipital cortex.
ETCo2 in mm Hg, to be recorded for the duration of the scan session and be synchronized with the single fMRI procedure timing
Visual Analog Scale (VAS) measurements of sleepiness, alertness, calm, tension, and anxiety performed before dosing (baseline), pre-fMRI session, post-fMRI session and just before leaving the facility.
Association between the anxiety trait (STAI-trait, test battery for neuroticism or liability for Anxiety Disorders) collected at screening and the various pharmacodynamic parameters measured in the various testing conditions.
GW876008 concentration to determine pharmacokinetic parameters to be collected twice per session,
Pharmacogenetic (PGx) assessments
Safety and tolerability of GW876008 to include Vital signs semi-supine; respiratory rate, pulse oximetry and ECG.
Clinical laboratory tests
fMRI BOLD ALS signal.
Heart rate (HR; beats per minute), to be recorded for the whole duration of the scan session and to be synchronized with the single fMRI procedure timing.
Respiratory rate (RR: inspiration per minute), to be recorded for the duration of scan session and be synchronized with the single fMRI procedure timing. .

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MBChB, MFPM, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, La Jolla, California, United States